CLINICAL TRIAL: NCT01006291
Title: A 26 Week Randomised, Controlled, Open Label, Multicentre, Multinational, Three-arm, Treat to Target Trial Comparing Efficacy and Safety of Three Different Dosing Regimens of Either Soluble Insulin Basal Analogue (SIBA) or Insulin Glargine With or Without Combination With OAD Treatment, in Subjects With Type 2 Diabetes Mellitus (BEGIN™ : FLEX)
Brief Title: Comparison of NN1250 With Insulin Glargine in Type 2 Diabetes
Acronym: BEGIN™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3668; U1111-1111-7084 (Other: WHO); 2008-005771-10 (EudraCT Number)
Record Dates: First submitted 2009-10-30; First posted 2009-11-02 (Estimated); Results first posted 2015-11-13 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2016-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IDeg OD FF (Experimental)
  Interventions: Drug: insulin degludec
- IDeg OD (Experimental)
  Interventions: Drug: insulin degludec
- IGlar OD (Experimental)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec — Injected s.c. (under the skin) once daily (alternative regimen). Dose was individually adjusted.
  Arms: IDeg OD FF
Drug: insulin degludec — Injected s.c. (under the skin) once daily. Dose was individually adjusted.
  Arms: IDeg OD
Drug: insulin glargine — Insulin glargine injected s.c. (under the skin) once daily. Dose was individually adjusted.
  Arms: IGlar OD

SUMMARY:
This trial is conducted in Africa, Asia, Europe and South America. The aim of this clinical trial is to compare NN1250 (insulin degludec (IDeg) with insulin glargine (IGlar) in patients with type 2 diabetes. Subjects treated with oral antidiabetic drug(s) (OAD(s)) should continue their current OAD treatment at the stable, prerandomisation dose level and dosing frequency.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (diagnosed clinically) for at least 6 months
* Current treatment: oral anti-diabetic drug(s) (OAD(s)) alone, basal insulin alone or the combination of OAD(s) and basal insulin. Allowed OADs are: Metformin, insulin secretagogues (sulphonylureas (SU) or glinides), pioglitazone with unchanged dosing for at least 3 months prior to Visit 1
* HbA1c: OADs only users 7.0-11.0 % (both inclusive), basal insulin with/without OADs users 7.0-10.0% (both inclusive) by central laboratory analysis
* Body Mass Index (BMI) below or equal to 40.0 kg/m^2

Exclusion Criteria:

* Cancer and medical history of cancer hereof
* Use within the last 3 months prior to Visit 1 of: glucagon-like peptide-1(GLP-1) receptor agonist (exenatide, liraglutide), rosiglitazone, dipeptidyl peptidase IV (DPP-IV) inhibitors, alpha-glucosidase-inhibitors
* Cardiovascular disease, within the last 6 months prior to Visit 1, defined as: stroke; decompensated heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Uncontrolled treated/untreated severe hypertension (systolic blood pressure at least 180 millimetre (mm) mercury (Hg) and/or diastolic blood pressure at least 100 mmHg)
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures according to local requirements
* Cancer and medical history of cancer hereof (except basal cell skin cancer and squamous cell skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 687 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (63):
- Argentina (3):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Ciudad Autónoma de Bs As
  - Novo Nordisk Investigational Site, Rosario
- Finland (6):
  - Novo Nordisk Investigational Site, Hanko
  - Novo Nordisk Investigational Site, Harjavalta
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Turku
  - Novo Nordisk Investigational Site, Vantaa
- Hungary (4):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Győr
  - Novo Nordisk Investigational Site, Szombathely
- India (10):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, New Dehli, New Delhi
  - Novo Nordisk Investigational Site, Chandigarh, Punjab
  - Novo Nordisk Investigational Site, Vellore, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Chennai
  - Novo Nordisk Investigational Site, Hyderabad
- Israel (8):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Jerusalem
  - Novo Nordisk Investigational Site, Kfar Saba
  - Novo Nordisk Investigational Site, Netanya
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Rehovot
- Malaysia (5):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, George Town
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
  - Novo Nordisk Investigational Site, Kuala Lumpur
  - Novo Nordisk Investigational Site, Putrajaya
- Mexico (3):
  - Novo Nordisk Investigational Site, Durango, Durango
  - Novo Nordisk Investigational Site, Mexico City, México, D.F.
  - Novo Nordisk Investigational Site, Monterrey
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Norway (6):
  - Novo Nordisk Investigational Site, Gjøvik
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Hønefoss
  - Novo Nordisk Investigational Site, Oslo
  - Novo Nordisk Investigational Site, Stavanger
  - Novo Nordisk Investigational Site, Tønsberg
- Russia (4):
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saint-Peterburg
- Novo Nordisk Investigational Site, Belgrade, Serbia
- South Africa (2):
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
- Taiwan (2):
  - Novo Nordisk Investigational Site, Taipei
  - Novo Nordisk Investigational Site, Taoyuan District
- United Kingdom (8):
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Edgbaston, Birmingham
  - Novo Nordisk Investigational Site, Edinburgh
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Hull
  - Novo Nordisk Investigational Site, Ipswich
  - Novo Nordisk Investigational Site, Londonderry
  - Novo Nordisk Investigational Site, Swansea

REFERENCES:
- [Result] Ratner RE, Gough SC, Mathieu C, Del Prato S, Bode B, Mersebach H, Endahl L, Zinman B. Hypoglycaemia risk with insulin degludec compared with insulin glargine in type 2 and type 1 diabetes: a pre-planned meta-analysis of phase 3 trials. Diabetes Obes Metab. 2013 Feb;15(2):175-84. doi: 10.1111/dom.12032. Epub 2012 Dec 3. PMID 23130654
- [Result] Sorli C, Warren M, Oyer D, Mersebach H, Johansen T, Gough SC. Elderly patients with diabetes experience a lower rate of nocturnal hypoglycaemia with insulin degludec than with insulin glargine: a meta-analysis of phase IIIa trials. Drugs Aging. 2013 Dec;30(12):1009-18. doi: 10.1007/s40266-013-0128-2. PMID 24170235
- [Result] Einhorn D, Handelsman Y, Bode BW, Endahl LA, Mersebach H, King AB. PATIENTS ACHIEVING GOOD GLYCEMIC CONTROL (HBA1c <7%) EXPERIENCE A LOWER RATE OF HYPOGLYCEMIA WITH INSULIN DEGLUDEC THAN WITH INSULIN GLARGINE: A META-ANALYSIS OF PHASE 3A TRIALS. Endocr Pract. 2015 Aug;21(8):917-26. doi: 10.4158/EP14523.OR. Epub 2015 Jun 29. PMID 26121451
- [Result] Russell-Jones D, Gall MA, Niemeyer M, Diamant M, Del Prato S. Insulin degludec results in lower rates of nocturnal hypoglycaemia and fasting plasma glucose vs. insulin glargine: A meta-analysis of seven clinical trials. Nutr Metab Cardiovasc Dis. 2015 Oct;25(10):898-905. doi: 10.1016/j.numecd.2015.06.005. Epub 2015 Jun 18. PMID 26232910
- [Result] Vora J, Seufert J, Solberg H, Kinduryte O, Johansen T, Hollander P. Insulin degludec does not increase antibody formation versus insulin glargine: an evaluation of phase IIIa trials. Diabetes Obes Metab. 2016 Jul;18(7):716-20. doi: 10.1111/dom.12621. Epub 2016 Feb 8. PMID 26663320
- [Derived] Meneghini L, Atkin SL, Gough SC, Raz I, Blonde L, Shestakova M, Bain S, Johansen T, Begtrup K, Birkeland KI; NN1250-3668 (BEGIN FLEX) Trial Investigators. The efficacy and safety of insulin degludec given in variable once-daily dosing intervals compared with insulin glargine and insulin degludec dosed at the same time daily: a 26-week, randomized, open-label, parallel-group, treat-to-target trial in individuals with type 2 diabetes. Diabetes Care. 2013 Apr;36(4):858-64. doi: 10.2337/dc12-1668. Epub 2013 Jan 22. PMID 23340894
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 69 sites in 14 countries: Hungary (3 sites), Macedonia (1 site), Serbia (3 sites), Finland (7 sites), Norway (6 sites), United Kingdom (6 sites), Argentina (4 sites), Mexico (2 sites), South Africa (3 sites), India (10 sites), Malaysia (5 sites), Taiwan (3 sites), Russian Federation (8 sites) and Israel (8 sites).
Groups:
- IDeg OD FF: Insulin degludec (IDeg) was given once daily (OD) subcutaneously (s.c.) with or without pre-trial OADs for 26 weeks with alternating morning and evening dosing according to a fixed flexible (FF) schedule (approximately 8-40 hours intervals between doses).
- IDeg OD: Insulin degludec (IDeg) was given once daily (OD) subcutaneously (s.c.) at main evening meal with or without pre-trial OADs for 26 weeks.
- IGlar OD: Insulin glargine (IGlar) was given once daily (OD) subcutaneously (s.c.) according to local labelling with or without pre-trial OADs for 26 weeks.
Period: Overall Study
Arm/Group | IDeg OD FF | IDeg OD | IGlar OD
Started | 229 | 228 | 230
Exposed | 230 (1 subject withdrew before exposure to drug. 2 subjects randomised to IDeg OD received IDeg OD FF) | 226 (2 subjects received IDeg OD FF) | 229 (1 subject withdrew prior to exposure to trial drug)
Completed | 203 | 204 | 203
Not Completed | 26 | 24 | 27
Not completed — Adverse Event | 2 | 1 | 2
Not completed — Lack of Efficacy | 2 | 2 | 1
Not completed — Protocol Violation | 3 | 3 | 3
Not completed — Withdrawal criteria | 5 | 4 | 4
Not completed — Other | 14 | 14 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg OD FF | IDeg OD | IGlar OD | Total
Number analyzed (Participants) | 229 | 228 | 230 | 687
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (10.3) | 56.5 (9.6) | 56.7 (8.8) | 56.4 (9.6)
Gender [Count of Participants; unit: Participants]
  Female | 94 | 104 | 119 | 317
  Male | 135 | 124 | 111 | 370
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.5 (1.0) | 8.4 (0.9) | 8.4 (0.9) | 8.4 (0.9)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.0 (2.6) | 8.8 (2.8) | 9.0 (2.8) | 8.9 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after 26 weeks of treatment
Time Frame: Week 0, Week 26
Population: The Full analysis set (FAS) included all randomised subjects and missing data is imputed using last observation carried forward (LOCF). In FAS, subjects contributed to the evaluation 'as randomised'.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDeg OD FF | IDeg OD | IGlar OD
Number analyzed (Participants) | 229 | 228 | 230
percentage of glycosylated haemoglobin | -1.28 (1.00) | -1.07 (0.99) | -1.26 (1.07)

2. Secondary Outcome: Mean of 9-point Self Measured Plasma Glucose Profile (SMPG)
Description: Mean of SMPG after 26 weeks of treatment. Plasma glucose measured: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, before bedtime, at 4 am and before breakfast.
Time Frame: Week 26
Population: The FAS included all randomised subjects and missing data is imputed using last observation carried forward (LOCF). In FAS, subjects contributed to the evaluation 'as randomised'. For 28 subjects all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg OD FF | IDeg OD | IGlar OD
Number analyzed (Participants) | 216 | 220 | 223
mmol/L | 7.9 (1.8) | 8.0 (2.1) | 7.8 (1.9)

3. Secondary Outcome: Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: The SAS included all subjects who received at least one dose of the investigational product or its comparator. In SAS, subjects contributed to the evaluation 'as treated'.230 subjects in the IDeg Flex group, 226 in the IDeg OD group and 229 in the IGlar OD group
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD FF | IDeg OD | IGlar OD
Number analyzed (Participants) | 230 | 226 | 229
Episodes/100 years of patient exposure | 364 | 363 | 348

4. Secondary Outcome: Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Rate of nocturnal confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes are defined as occurring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: as for outcome 3
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDeg OD FF | IDeg OD | IGlar OD
Number analyzed (Participants) | 230 | 226 | 229
Episodes/100 years of patient exposure | 63 | 56 | 75

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 26 weeks + 7 days follow up
Description: Safety analysis set includes all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDeg OD FF | IDeg OD | IGlar OD
Serious Adverse Events (participants affected / at risk) | 6/230 | 8/226 | 4/229
Other Adverse Events (participants affected / at risk) | 58/230 | 57/226 | 53/229
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD FF (N=230) | IDeg OD (N=226) | IGlar OD (N=229)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Oral neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Transurethral prostatectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg OD FF (N=230) | IDeg OD (N=226) | IGlar OD (N=229)
Diarrhoea (Gastrointestinal disorders) | 10 (12) | 14 (17) | 10 (11)
Nasopharyngitis (Infections and infestations) | 23 (28) | 20 (28) | 18 (21)
Upper respiratory tract infection (Infections and infestations) | 20 (21) | 11 (14) | 20 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (13) | 9 (9) | 6 (9)
Dizziness (Nervous system disorders) | 3 (3) | 3 (3) | 12 (13)
Headache (Nervous system disorders) | 16 (25) | 16 (18) | 9 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.